CLINICAL TRIAL: NCT05651737
Title: Efficacy of an Unguided or Peer-guided App-based Psychosocial Intervention to Enhance Quality of Life in Arabic-speaking Refugees Residing in Switzerland: A Randomized Controlled Trial
Brief Title: App-based Psychosocial Intervention to Enhance Quality of Life in Arabic-speaking Refugees Residing in Switzerland
Acronym: Sui
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss Transfusion SRC (Other); Freie Universität Berlin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-00607
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Quality of Life; Stigma, Social; Depression; PTSD; Anxiety
MeSH Terms: conditions — Social Stigma; Depression; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sui App+ (peer guided) (Active Comparator): The active phase of the study is eight weeks per participant with a follow-up online assessment after another eight weeks.
  One of the active study groups, the Sui App+ condition, receives the Sui app plus a peer who will guide them online. They receive weekly individual messages from their peer within the chat of the app.
  Interventions: Behavioral: Sui App (SRK)
- Sui App (unguided) (Active Comparator): The active phase of the study is eight weeks per participant with a follow-up online assessment after another eight weeks.
  The second active study group receives the app as a standalone intervention. They use whatever content they are interested in and receive weekly push-notifications in case they were not active.
  Interventions: Behavioral: Sui App (SRK)
- Waitlist control group (No Intervention): The control arm is a waitlist control group that receives access to the app after eight weeks.

INTERVENTIONS:
Behavioral: Sui App (SRK) — The Sui app contains the following chapters:
  6 well-being chapters on: stress, sleep, resources throughout the day, chronic pain, emotion regulation, audio exercises 9 Swiss-specific information chapters on: housing, health (two sub-chapters), finances, asylum process, residence status, social integration, occupational integration, family reunification
  Arms: Sui App (unguided); Sui App+ (peer guided)

SUMMARY:
The ongoing warfare and economic instability in the Middle East and in North Africa causes many people to leave their home countries. Arrived in a host countries, in this example, in Switzerland, they face a lot of structural and psychosocial hurdles. Particularly in the first years, building up a certain quality of life is complicated and challenging. To support this process, the Swiss Red Cross and the University of Bern have developed the Sui app. It contains structural and social information as well as low-intensity psychological tools to provide support to the everyday life of Arabic-speaking people in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Arabic as native or second language
* Good knowledge of reading, writing and speaking Arabic
* Have lived in Switzerland for no longer than 5 years
* Give written consent
* Have access to a smartphone and an internet connection
* Indicate an emergency contact whom they could contact in event of a crisis

Exclusion Criteria:

* Indicate an increased risk of self-harm or suicide at baseline
* Indicate having been diagnosed with psychosis or bipolar disorder
* Be participating in a similar study at baseline
* Have a lack of written and spoken Arabic skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Well-being at baseline | Baseline
  Measured by the WHO Quality of Life Short Version (WHOQOL-BREF, 4 domain scores, mean score multiplied by 4, 0 (low) to 100 (high) range)
Well-being at post-intervention timepoint | Post (after 8 weeks)
  Measured by the WHO Quality of Life Short Version (WHOQOL-BREF, 4 domain scores, mean score multiplied by 4, 0 (low) to 100 (high) range)
Well-being at follow-up timepoint | Follow-Up (after 16 weeks)
  Measured by the WHO Quality of Life Short Version (WHOQOL-BREF, 4 domain scores, mean score multiplied by 4, 0 (low) to100 (high) range)

SECONDARY OUTCOMES:
Satisfaction with the treatment | Post (after 8 weeks), Follow-Up (after 16 weeks)
  Measured by the Questionnaire on satisfaction with the treatment (ZUF-8, 1(low) to 4 (high) scores) adapted for "app" as intervention
Self-stigma | Baseline, Post (after 8 weeks), Follow-Up (after 16 weeks)
  Measured by the Self-stigma of mental illness scale short form (SSMIS-SF, 1(strongly disagree) to 9 (strongly agree) scores)
PTSD symptoms | Baseline, Post (after 8 weeks), Follow-Up (after 16 weeks)
  Measured by the Post traumatic stress disorder checklist scale according to DSM-5 (PCL-5, 0 (not at all) to 80 (extremely) range)
Somatic symptoms | Baseline, Post (after 8 weeks), Follow-Up (after 16 weeks)
  Measured by the Patient Health Questionnaire 15 (PHQ-15, 0 (normal) to 30 (severe) symptom range )
Anxiety symptoms | Baseline, Post (after 8 weeks), Follow-Up (after 16 weeks)
  Measured by the Generalised Anxiety Disorder 7 (GAD-7, 0 (minimal) to 21 (severe) symptom range)
Depressive symptoms | Baseline, Post (after 8 weeks), Follow-Up (after 16 weeks)
  Measured by the Patient Health Questionnaire 9 (PHQ-9, 0 (no suspicion of) to 27 (suspicion of severe) depression range)
Post migration stressors | Baseline, Post (after 8 weeks), Follow-Up (after 16 weeks)
  Measured by the Post-migratory life difficulties Checklist (PMLD-CL, 0 (no) to 4 (very serious) post migration problem scores)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berger, Prof. Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No